CLINICAL TRIAL: NCT06872814
Title: Vaccine Hesitancy in Patients with Solid Tumors: a Cross-sectional Single-center Survey
Acronym: VE
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Angioletta Lasagna, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: VE
Record Dates: First submitted 2025-03-07; First posted 2025-03-12 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-02

CONDITIONS: Cancer Patients; Vaccine-Preventable Diseases
MeSH Terms: conditions — Vaccine-Preventable Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
Cancer patients have a well-known and higher risk of vaccine-preventable disease (VPD) than the general population. VPD can cause serious complications due to compromised immune system, malnutrition and the same oncology treatments and represent a severe financial burden with a delay in treating the underlying cancer The main purpose of this survey is to analyse the perception of cancer patients on the topic vaccines and vaccine-preventable diseases, the acceptability of vaccines and the evaluation of the determining factors associated with the choice of the patient to be vaccinated or not. This information will be used to improve the management of these issues.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years of age;
2. Oncology patient defined as a patient with solid tumors undergoing active systemic treatment or follow-up;
3. Written informed consent

Exclusion Criteria:

1. Patients with hematological tumors
2. Patients who are unable to understand informed consent document

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of this cross-sectional survey will include out-patients of the Medical Oncology Unit, Fondazione IRCCS Policlinico San Matteo Pavia
Sampling Method: Non-Probability Sample
Enrollment: 309 (Actual)
Dates: Start 2024-05-31 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2024-08-26 (Actual)

PRIMARY OUTCOMES:
assess the proportion of vaccinated subjects in our cohort of cancer patients undergoing active cancer treatment | 3 months
  The primary endpoint will be to assess the proportion of vaccinated subjects in the investigators cohort of cancer patients undergoing active cancer treatment (number of patients who received at least one vaccine/ total number of patients)

SECONDARY OUTCOMES:
assess the proportion of vaccinated subjects with the anti flu vaccine in the investigators cohort of cancer patients undergoing active cancer treatment | 3 months
assess the proportion of vaccinated subjects with anti SARS-CoV-2 vaccine in the investigators cohort of cancer patients undergoing active cancer treatment | 3 months
assess the proportion of vaccinated subjects with anti pneumococccal vaccine in the investigators cohort of cancer patients undergoing active cancer treatment | 3 months
assess the proportion of vaccinated subjects with anti HZ vaccine in the investigators cohort of cancer patients undergoing active cancer treatment | 3 months
assess which variables (sex, age, degree of education, marital state, commodities, type of tumor, type of oncological treatment) are associated with not willingness to receive vaccines | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, SC Oncologia, Pavia, Pavia, Italy